CLINICAL TRIAL: NCT03944499
Title: A Phase I,Multicenter,Open-label,Single-arm Study:A Dose-escalation Phase Evaluating FS1502 in Patients With HER2 Expressed Advanced Solid Tumors,and a Dose-expanded Phase in Patients With Local Advanced or Metastatic,HER2+ Breast Cancer
Brief Title: Phase 1 Study of FS-1502 in Patients With HER2 Expressed Advanced Solid Tumors and Breast Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS-CY1502-Ph1-01
Record Dates: First submitted 2019-04-30; First posted 2019-05-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FS-1502 (Experimental): Phase Ia:
  Patients enrolled on the 1.2 and 2.0 regimens: FS-1502 monotherapy every 4 weeks with intravenous drip, 28 days as a cycle; Patients enrolled on the 3.0 regimens: starting from the 1.0mg/kg dose group, FS-1502 monotherapy every 3 weeks with intravenous drip, 21 days as a cycle;
  Phase Ib:
  FS-1502 monotherapy, the dose and frequency of administration for Stage Ib will be obtained according to Phase Ia (RP2D). All patients will continue treatment until no clinical benefit occurs, or intolerable toxicity occurs, or death occurs, or the investigator decides, or patients voluntarily withdraw from the study.
  Study end is defined as the last patient's treatment ended or 2 years after the last patient's treatment began(depending on which happens earlier).
  Interventions: Drug: FS-1502

INTERVENTIONS:
Drug: FS-1502 — Dose-Escalation Phase (Phase 1a)： FS-1502 dose-escalation will be proceeded on standard 3+3 design with starting dose of 0.1 mg/kg, IV, once per 28 days, 28 days as a cycle in the V1.2 and V2.0 regimens; IV, once per 21 days, 21 days as a cycle in the V3.0 regimens..
  Dose level 1: 0.1 mg/kg; Dose level 2: 0.2 mg/kg; Dose level 3: 0.4 mg/kg; Dose level 4: 0.6 mg/kg; Dose level 5: 0.8 mg/kg; Dose level 6: 1.0 mg/kg; Dose level 7: 1.3 mg/kg. If 1.3mg/kg is still tolerated safely and in line with linear kinetic characteristics, and combined with the results of PK, PD, safety and effectiveness, a comprehensive assessment is made to determine whether to continue the dose escalating. The subsequent dose increase ratio is 33% (the dose increase ratio can be adjusted according to the previous data results) until MTD or RP2D.
  Dose-expansion Phase (Phase 1b) : RP2D determined in phase 1a, IV.

SUMMARY:
The study comprises two phases: Phase 1a and Phase 1b. The purpose of the study is to observe the safety， tolerability and efficacy of FS-1502.

DETAILED DESCRIPTION:
The study is designed as an open label, single arm, Phase 1a/1b study with a dose-escalation phase to evaluate FS-1502 in patients with HER2 expressed advanced malignant solid tumors (phase 1a) and an expanded cohort (phase 1b) to evaluate FS-1502 in patients with metastatic, HER2-positive breast cancer. The primary aim of the phase 1a portion of this study is to determine the safety and tolerability of FS-1502. The primary aim of the phase 1b portion is to demonstrate efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study registration (men and women eligible);
2. Phase Ia dose-escalation study:

   Patients with HER2-expressing advanced malignant solid tumors who had failed to standard therapy(including surgery, chemotherapy, radiation therapy or biotherapy) , or can not receive standard therapy, or no standard therapy is available.
   1. HER2 expression: IHC3+, IHC2+/FISH+
   2. HER2 expression: IHC1+, IHC2+/FISH-

   Phase Ib dose-expanded study:

   Histologically or cytologically confirmed HER2-positive patients with advanced breast cancer who had previously received at least 2 line therapy and had failed anti-HER2 therapy. Details as follows:
   1. HER2 positive (defined as IHC3+ or IHC2+/FISH+);
   2. For patients with advanced breast cancer who had previously failed anti-HER2 therapy and had received at least 2-line therapy, postoperative adjuvant therapy which could be considered as a treatment line number if disease progression during treatment and within 12 months after completion of treatment.
   3. Provide evidence of disease progression or intolerable toxicity as confirmed by the investigator or medical history recorded prior to enrollment.
   4. The enrollment can be based on written HER2 test report from certified local lab, and if patients had no HER2 test report, they should provide sufficient paraffin sections or fresh tumor tissue specimens which should be sent to the local lab or the central laboratory for testing and confirmation.

   Pivotal clinical study:

   Patients with locally advanced or relapsed metastatic breast cancer who have been histologically or cytologically confirmed to be HER2-positive and who have received two or more lines of anti-HER2 therapy in the past. Details as follows:
   1. Her2-positive patients: Patients with IHC3+ or IHC2+ and FISH positive patients should provide enough tumor tissue samples within 5 years for the central laboratory to confirm HER2 status. Patients with HER2-positive patients are considered to be eligible for inclusion in this study; If the specimens provided are undetectable or are not available, a positive HER2 test from a local laboratory approved by the NMPA may be reported for entrainment.
   2. Previous treatment with two or more lines of anti-HER2 therapy, neoadjuvant therapy or adjuvant therapy can be used as a treatment line number if the disease progresses during or within 12 months after treatment.
   3. Evidence of investigator-confirmed or documented disease progression or intolerance of toxicity prior to enrollment.
3. The ECOG performance status must be 0 or 1.
4. Expected survival for at least 12 weeks.
5. Has adequate organ and bone marrow function: absolute neutrophil count (ANC) ≥ 1.0x1E9/L(without colony stimulating factor within 7 days); hemoglobin ≥ 90g/L (without red blood cell infusion within 14 days); platelet count ≥ 100x1E9/L(without thrombopoietin or thrombopoietin receptor agonists within 7 days nor platelet infusion within 14 days); Total bilirubin ≤ 1.5x upper limit normal (ULN), or ≤ 3x ULN if with Gilbert syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN; AST and ALT ≤ 5x ULN if liver metastasis; Serum creatinine < 1.5x ULN and creatinine clearance ≥ 50mL/min (Cockroft-Gault formula calculation); Serum potassium ≥3.5 mmol/L；albumin ≥ 3g/dL; left ventricular ejection fraction (LVEF) >50%；urinary protein ≤1+ or 24-hour urinary protein dose < 1.0g.
6. Has at least one non-intracranial measurable lesion by RECIST version 1.1.
7. Male or female patients with fertility must agree to use effective contraceptive methods during the study period and within 3 months of the last dose of study therapy, such as dual barrier contraceptive methods, condoms, oral or injectable contraceptives, and intrauterine devices.
8. Ability to understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. Patients who received chemotherapy, targeted therapy, radiotherapy, etc., 14 days or within 5 half-lives periods, whichever is shorter, prior to the start of dosing. Patients who received major surgery, tumor immunotherapy, or monoclonal antitumor therapy within 4 weeks prior to the start of dosing.
2. Patients who have participated in other clinical trials 4 weeks before the start of study drug administration or within 5 half-lives periods, whichever is shorter.
3. Patients previously treated with anti-HER2 ADC drugs.
4. Patients with central nervous system metastasis.
5. Clinically uncontrolled mass pleural effusion, pericardial effusion, or abdominal effusion (2 weeks before first administration).
6. Non-recovery of toxic effects from previous antitumor therapy (> NCI-CTCAE 5.0 grade 1) alopecia, neurotoxicity, or other toxicity that had become chronic as assessed by the investigator and did not affect the safety of the investigational medication was admitted to NCI-CTCAE 5.0 grade 2 or below.
7. Patients with corneal epitheliopathy (other than mild punctiform keratopathy or existing eye diseases affecting the evaluation of ocular toxicity after trial administration) or who were unwilling to stop wearing contact lenses during the study.
8. Patients take medications that prolong the QTc interval (mainly Ia, Ic, Class III antiarrhythmic drugs) or have risk factors that prolong the QTc interval, such as uncorrectable hypokalemia, hereditary long QT syndrome;
9. Cardiac function and disease conform to one of the following conditions:

   1. Three 12-lead electrocardiogram (ECG) measurements were performed at the research center during the screening period, and three mean values were calculated according to the QTc formula adopted by the instrument, QTc > 470 ms;
   2. New York Heart Association (NYHA)Grade ≥ 2 for congestive heart failure;
   3. arrhythmia of clinical significance grade ≥ 2.
   4. History of myocardial infarction or severe arteriovenous thrombosis within 6 months.
10. Pregnant or lactating women;
11. Known allergy to any excipients of FS-1502;
12. Active infections requiring systemic treatment;
13. Persons with active hepatitis B (HBV surface antigen positive with HBV DNA exceeding 1000 IU/ml or meeting the research Center criteria for diagnosis of active hepatitis B infection) or hepatitis C (HCV RNA positive), human immunodeficiency virus infection (HIV positive);
14. Had been diagnosed with any other malignancies within the 5 years prior to study participation, other than early malignancies that have undergone radical treatment (carcinoma in situ), such as adequately treated basal or squamous cell skin cancers or carcinoma in situ of the cervix;
15. Any other clinically significant disease or condition that the investigator believes may affect protocol compliance or affect the patient's signing of the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
DLT of first single dose of FS-1502. | At the end of Cycle 1 (each cycle is 28 days or 21 days) in Phase Ia.
  DLT is defined as a dose-limiting toxicity event occurring during the DLT observation period that, as determined by the Investigator and/or Sponsor to be at least possibly related to FS-1502, is classified using NCI-CTCAE version 5.0 as conforming to AE or laboratory anomalies specified in the protocol.
MTD of single dose of FS-1502 | At the end of Cycle 1 (each cycle is 28 days or 21 days) in Phase Ia.
  MTD was defined as the maximum dose of < 33% DLT events observed in patients with evaluable DLT events (i.e., 1 in 6 patients at most or 0 in 3 patients).
Recommend Phase 2 Dose(RP2D) of single dose of FS-1502 | Throughout the Phase Ia
  If the MTD is not observed, the appropriate therapeutic exposure dose or RP2D is determined based on the antitumor efficacy evaluation, safety data, and PK data.
Overall response rate (ORR) assessed by IRC | Approximately 2 years in Phase Ib.
  Percentage of patients with confirmed CR or PR as evaluated by RECIST version 1.1

SECONDARY OUTCOMES:
TEAE | Approximately 3 years.
  Incidence Rate and type of treatment emergent adverse event that were evaluated according to CTCAE version 5.0.
SAE and AE that leading to treatment permanent discontinuation | Approximately 2 years.
  Number of Participants with serious adverse events and adverse reactions that leading to treatment permanent discontinuation of FS1502.
Incidence of deaths and causes | Approximately 3 years.
  Incidence of deaths and causes within 30 days after the last dose.
Progression free survival (PFS) | Approximately 2 years.
  Progression free survival is defined as the time from the beginning of randomization until disease progression or death, whichever occurred first.For patients without an event (no progression or death), the cut-off point will be the date of the last tumor evaluation.For patients without an evaluation of efficacy after baseline, the cut-off point was the first dosing date.
Overall survival (OS) | Approximately 3 years.
  Overall survival is defined as the time from randomization to death from any cause.For patients with no observed death events, the cut-off point will be the date of the last time patient survival information was obtained.
1-year overall survival (OS) rate | 1 years
  1-year overall survival (OS) rate is defined as the proportion of patients who survived 1 year after the initiation of randomization.
Duration of response (DoR) | 2 years
  Duration of response is defined as the time from the first CR or PR to tumor progression or death from any cause, whichever occurs first.If there is no tumor progression or death, the cut-off point will be the date of the last tumor evaluation.
Clinical benefit response (CBR) | Approximately 2 years
  Percentage of participants achieve clinical benefit (complete response (CR), partial response (PR) or stable disease (SD) more than 6 months) from the treatment.
Area under the serum concentration versus time curve (AUC) | Approximately 2 years.
  Measure the AUC of FS-1502 and it metabolites (MMAF).
Peak Serum Concentration (Cmax) | Approximately 2 years.
  Measure the Cmax of FS-1502 and it metabolites (MMAF).
Time to maximum concentration (tmax) | Approximately 2 years.
  Measure the tmax of FS-1502 and it metabolites (MMAF).
Elimination half life (T1/2) | Approximately 2 years.
  Measure the T1/2 of FS-1502 and it metabolites (MMAF).
Clearance (Cl) | Approximately 2 years.
  Measure the Clearance of FS-1502 and it metabolites (MMAF).
Anti-FS-1502 antibody | Approximately 2 years.
  Measure the anti-FS-1502 antibody to demonstrade the immunogenicity of FS-1502.

CONTACTS AND LOCATIONS:
Overall Officials: BINGHE XU, PhD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (12):
- China (12):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Jilin, Changchun
  - Sun Yat-sen University Cancer Prevention Center, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shenzhen Hospital, Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Run Run Shaw Hospital Affiliated to Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No